CLINICAL TRIAL: NCT02319837
Title: A Phase 3, Randomized, Efficacy and Safety Study of Enzalutamide Plus Leuprolide, Enzalutamide Monotherapy, and Placebo Plus Leuprolide in Men With High-Risk Nonmetastatic Prostate Cancer Progressing After Definitive Therapy
Brief Title: Safety and Efficacy Study of Enzalutamide Plus Leuprolide in Patients With Nonmetastatic Prostate Cancer (EMBARK)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-13; C3431004 (Other: Alias Study Number); 2024-513521-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2014-12-14; First posted 2014-12-18 (Estimated); Results first posted 2024-03-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Hormone Sensitive Prostate Cancer; Prostate Cancer; Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; luprolide acetate gel depot; Leuprolide

STUDY DESIGN:
Masking Description: The randomized blinded portion of the study has concluded. The study is now being conducted open label manner.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enzalutamide plus leuprolide (Experimental): Enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily in combination with leuprolide administered as as a single intramuscular or subcutaneous injection once every 12 weeks
  Interventions: Drug: Enzalutamide; Drug: Leuprolide Open Label
- Enzalutamide monotherapy (Experimental): Enzalutamide (160 mg) administered as four 40-mg capsules by mouth once daily
  Interventions: Drug: Enzalutamide
- Leuprolide plus placebo (Active Comparator): Enzalutamide placebo (placebo) capsules (identical in appearance to enzalutamide) administered as 4 capsules by mouth once daily in combination with leuprolide administered as a single intramuscular or subcutaneous injection once every 12 weeks.
  The randomized blinded portion of the study has concluded following primary endpoint analyses. In the Open Label Period the placebo is no longer applicable in this study arm, and patients continue to receive leuprolide alone.
  Interventions: Drug: Placebo (No longer applicable in Open Label study period)

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: MDV3100; Xtandi
  Arms: Enzalutamide monotherapy; Enzalutamide plus leuprolide
Drug: Placebo (No longer applicable in Open Label study period) — Sugar pill to mimic enzalutamide
  Arms: Leuprolide plus placebo
Drug: Leuprolide Open Label
  Other Names: Eligard; Leuprolide Acetate; Leuprorelin; Lupron
  Arms: Enzalutamide plus leuprolide

SUMMARY:
The purpose of this study is to assess enzalutamide plus leuprolide in patients with high-risk nonmetastatic prostate cancer progressing after radical prostatectomy or radiotherapy or both.

The randomized / blinded portion of the study is now completed following primary endpoint analyses. The study remains ongoing in open label format.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate at initial biopsy, without neuroendocrine differentiation, signet cell, or small cell features;
* Prostate cancer initially treated by radical prostatectomy or radiotherapy (including brachytherapy) or both, with curative intent;
* PSA doubling time ≤ 9 months;
* Screening PSA by the central laboratory ≥ 1 ng/mL for patients who had radical prostatectomy (with or without radiotherapy) as primary treatment for prostate cancer and at least 2 ng/mL above the nadir for patients who had radiotherapy only as primary treatment for prostate cancer;
* Serum testosterone ≥ 150 ng/dL (5.2 nmol/L).

Exclusion Criteria:

* Prior or present evidence of distant metastatic disease as assessed by radiographic imaging;
* Prior hormonal therapy. Neoadjuvant/adjuvant therapy to treat prostate cancer ≤ 36 months in duration and ≥ 9 months before randomization, or a single dose or a short course (≤ 6 months) of hormonal therapy given for rising PSA ≥ 9 months before randomization is allowed.;
* Prior cytotoxic chemotherapy, aminoglutethimide, ketoconazole, abiraterone acetate, or enzalutamide for prostate cancer;
* Prior systemic biologic therapy, including immunotherapy, for prostate cancer;
* Major surgery within 4 weeks before randomization;
* Treatment with 5-α reductase inhibitors (finasteride, dutasteride) within 4 weeks of randomization;
* Known or suspected brain metastasis or active leptomeningeal disease;
* History of another invasive cancer within 3 years before screening, with the exception of fully treated cancers with a remote probability of recurrence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1068 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2026-09-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (244):
- United States (70):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - Cedars-Senai OCC Pharmacy, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sutter Medical Group, Vascular & Varicose Vein Center, Roseville, California
  - Sutter Medical Group, Roseville, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California, Davis, School of Medicine, Sacramento, California
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology, P.C., Golden, Colorado
  - Eastern Connecticut Hematology Oncology Associates, Norwich, Connecticut
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - First Urology, PSC, Jeffersonville, Indiana
  - The University of Kansas Hospital, Kansas City, Kansas
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - GU Research Network/Wichita Urology Group, Wichita, Kansas
  - John Hopkins University Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Sidney Kimmel Cancer Center at Johns Hopkins Hospital- Oncology Investigational Drug Services, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Comprehensive Urology - Macomb Office, Macomb, Michigan
  - Comprehensive Urology - Royal Oak (Stephenson) office, Royal Oak, Michigan
  - GU Research Network, LLC / Urology Cancer Center, Omaha, Nebraska
  - VA Lahontan Valley Outpatient Clinic, Fallon, Nevada
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center Westchester, Harrison, New York
  - Memorial Hospital, New York, New York
  - Sidney Kimmel Center for Prostate and Urologic Cancers, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Memorial Sloan Kettering Cancer Center Rockville Centre, Rockville Centre, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Memorial Sloan Kettering Cancer Center Nassau, Uniondale, New York
  - Duke Investigational Chemotherapy Services, Durham, North Carolina
  - Duke Nuclear Medicine, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - TriState Urologic Services PSC Inc., dba The Urology Group, Cincinnati, Ohio
  - Mercy Health Jewish Hospital, Cincinnati, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Southwest Urology, Middleburg Heights, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Imaging Center, Eugene, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - Honickman Centre, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Bodine Buiding, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Medical Oncology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt Unversity Medical Center, Dept. of Urologic Surgery, Nashville, Tennessee
  - Vanderbilt Unversity Medical Center, The Urology Clinic, Nashville, Tennessee
  - Urology Clinics of North Texas, PLLC, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Henrico Doctor's Hospital, Henrico, Virginia
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLLC., Virginia Beach, Virginia
- Australia (26):
  - Genesis Cancer Care NSW, Gateshead, New South Wales
  - Lismore Base hospital, Lismore, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Genesis Cancer Care, North Sydney, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Australian Clinical Trials Pty Ltd, Wahroonga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Crown Princess Mary Cancer Centre, Westmead, NEW
  - Icon Cancer Care Wesley, Auchenflower, Queensland
  - Icon Cancer Care Chermside, Chermside, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Icon Cancer Centre Southport, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Australian Urology Associates, Malvern, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (8):
  - Hospital Barmherzige Schwestern Linz, Linz, Upper Austria
  - Hospital Barmherzige Schwestern Linz, Department of Urology, Linz
  - Ordensklinikum Linz GmbH, Linz
  - Department of Nuclear Medicine and Endocrinology, University Hospital Salzburg, Austria, Salzburg
  - Department of Radiology, University Hospital Salzburg, Austria, Salzburg
  - Department of Urology,Paracelsus Medical University Salzburg, Salzburg
  - AKH - Medizinische Universität Wien, Vienna
  - Department of Internal Medicine I, Medical university Vienna, Vienna
- Brazil (10):
  - Hospital São Rafael S.A, Salvador, Estado de Bahia
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - CITO - Centro Integrado de Terapia Onco-Hematologica - Hospital de Clinicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CLINIONCO - Clinica de Oncologia de Porto Alegre Ltda., Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital das Clinicas da Faculdade de Ciencias Medicas da UNICAMP, Campinas, São Paulo
  - Centro de Estudos e Pesquisas de Hematologia e Oncologia - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Oncosite - Centro de Pesquisa Clinica em Oncologia Ltda, Ijuí/RS
- Canada (19):
  - Prostate Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Manitoba Prostate Centre CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - The Male/Female Health and Research Centre, Royal Court Medical Centre, Barrie, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - Urology Associates/ Urologic Medical Research, Kitchener, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Ultra-Med Inc., Pointe-Claire, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec - CRCEO, Québec, Quebec
- Denmark (6):
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen N, Copenhagen N
  - Aarhus University Hospital, Arhus N
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
  - Rigshospitalet, Dept of Radiology, Copenhagen
  - Odense University Hospital, Odense C
  - Vejle Sygehus, Vejle
- Finland (5):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Oulun yliopistollinen sairaala, Oulu
  - Satakunnan Keskussairaala, Pori
  - Seinaejoen Keskussairaala, Seinäjoki
  - Tampereen yliopistollinen sairaala, Tampere
- France (14):
  - ICO- site Paul Papin, Angers
  - Clinique Pasteur - Lanroze Service Pharmacie, Brest
  - Clinique Pasteur - Lanroze, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - ICM Val d'Aurelle, Montpellier
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHP Saint-Gregoire, Saint-Grégoire
  - ICO - site Rene Gauducheau, Saint-Herblain
  - Hia Begin, Saint-Mandé
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Italy (22):
  - Farmacia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Struttura Complessa di Oncologia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - UO di Radiologia, Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - UO di Oncologia,Ospedale Civile degli Infermi, Faenza RA
  - UO di Radiologia, Ospedale Civile degli Infermi, Faenza RA
  - UO di Oncologia, Ospedale Civile Umberto I, Lugo RA
  - Uo di Radiologia, Ospedale Civile Umberto I, Lugo RA
  - Laboratorio Farmaci Antiblastici, IRCCS Istituto, Meldola (FC)
  - U.O. Oncologia Medica, IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola (FC)
  - UO Radiologia,IRCCS Istituto Scientifico Romagnolo Per lO Studio e la Cura dei Tumori (IRST), Meldola (FC)
  - Istituto Nazionale Tumori Fondazione G. Pascale/Oncologia Medica A, Napoli
  - S.C.D.U. Oncologia Medica, A.O.U. San Luigi Gonzaga, Orbassano (TO)
  - S.C.D.U. Radiodiagnostica, A.O.U. San Luigi Gonzaga, Orbassano (TO)
  - Servizio di Farmacia, Ospedale Santa Maria delle Croci, Ravenna
  - Servizio di Radiologia, Ospedale Santa Maria Delle Croci, Ravenna
  - UO di Oncologia Medica, Ospedale Santa Maria delle Croci, Ravenna
  - Farmacia Interna, Ospedale degli Infermi, Rimini
  - UO Oncologia, Ospedale degli Infermi, Rimini
  - Azienda Ospedaliera S, Camillo Forlanini, UOC per il governo clinico in Oncologia Medica,pad,Flajani, Roma
  - U.O. di Oncologia Medica, Ospedale Santa Chiara, Trento
  - U.O. Medicina Nucleare, Ospedale Santa Chiara, Trento
  - U.O. Radiologia, Ospedale Santa Chiara, Trento
- Netherlands (8):
  - VU Medical Centrum, Department of Urology, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Gelderse Vallei Ziekenhuis, Ede
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - University Medical Centrum Groningen, Department Urologie, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht University Medical Center, Department of Urology, Maastricht
  - Antonius Ziekenhuis, Sneek
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii i Radioterapii, Gdansk
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o. o., Słupsk
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Oddzial Urologiczny, Słupsk
  - Kujawsko-Pomorskie Centrum Urologicznw Sp z o.o, Torun
  - Centrum Medyczne Melita Medical, Wroclaw
  - EMC Instytut Medyczny Spolka Akcyjna, Wroclaw
- Slovakia (7):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta, Banská Bystrica
  - CUIMED, s.r.o., Urologicka ambulancia, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - Univerzitna nemocnica Martin, Martin
  - UROEXAM, spol. s r.o., Nitra
  - MILAB, Prešov
  - Fakultna nemocnica s poliklinikou Zilina, Žilina
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital. Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, LA Coruna
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Dr. Antonio Alcaraz Asensio, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - ICO Girona; Hospital Universitari de Girona Dr. Josep Trueta. Servicio de Oncologia, Girona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon. Servicio de Oncologia., Madrid
  - Centro Oncologico MD Anderson International Espana, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Instituto Valenciano de Oncologia IVO, Valencia
- Sweden (7):
  - Sahlgrenska Universitetssjukhuset, Sahlgrenska, Gothenburg
  - Skanes Universitetssjukhus, Malmo
  - Universitetssjukhuset Orebro, Örebro
  - Sodersjukhuset AB, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (7):
  - Ross Hall Hospital, Glasgow, CITY of Glasgow
  - Royal Devon & Exeter Hospital, Wonford, Devon
  - Royal Free Hospital, London, Greater London
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Cancer Centre, Queen Elizabeth Hospital, Birmingham, WEST Midlands
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shore ND, Gleave M, De Giorgi U, Rannikko A, Pieczonka CM, Sridharan S, Brasso K, Woo HH, Gomez Caamano A, Saranchuk JW, Nordquist LT, Ferreira U, Tang Y, Rosbrook B, Haas GP, Rosales M, Zohren F, Tarazi J, Freedland SJ. Treatment of High-Risk Biochemically Recurrent Prostate Cancer With Enzalutamide in Combination With Leuprolide: Secondary Endpoints From the EMBARK Trial. J Urol. 2025 Dec 9:101097JU0000000000004890. doi: 10.1097/JU.0000000000004890. Online ahead of print. PMID 41364813
- [Derived] Shore ND, De Giorgi U, Tutrone RF, Bailen JL, Roos EPM, Kliment J, Marx G, Karsh LI, Ramirez-Backhaus M, Uchio EM, Supiot S, Tang Y, Rosbrook B, Haas GP, Rosales M, Zohren F, Tarazi J, Freedland SJ. Enzalutamide Monotherapy for the Treatment of Prostate Cancer With High-Risk Biochemical Recurrence: EMBARK Secondary End Points. J Urol. 2025 Dec 17:101097JU0000000000004879. doi: 10.1097/JU.0000000000004879. Online ahead of print. PMID 41349040
- [Derived] Shore ND, Luz MA, De Giorgi U, Gleave M, Gotto GT, Pieczonka CM, Haas GP, Kim CS, Ramirez-Backhaus M, Rannikko A, Kalac M, Sridharan S, Rosales M, Tang Y, Tutrone RF Jr, Venugopal B, Villers A, Woo HH, Wang F, Freedland SJ. Improved Survival with Enzalutamide in Biochemically Recurrent Prostate Cancer. N Engl J Med. 2025 Oct 19. doi: 10.1056/NEJMoa2510310. Online ahead of print. PMID 41124201
- [Derived] De Giorgi U, Freedland SJ, Rannikko A, Ramirez-Backhaus M, Villers A, Tarazi J, Tang Y, Haas GP, Rosales M, Shore ND. Enzalutamide in patients with high-risk biochemically recurrent prostate cancer according to the European Association of Urology definition: a post hoc analysis of EMBARK. Prostate Cancer Prostatic Dis. 2025 Mar 26. doi: 10.1038/s41391-025-00959-8. Online ahead of print. PMID 40140551
- [Derived] Freedland SJ, Gleave M, De Giorgi U, Rannikko A, Pieczonka CM, Tutrone RF, Venugopal B, Woo HH, Ramirez-Backhaus M, Supiot S, Lantz A, Ganguli A, Ivanova J, Kral P, Huang SP, Saad F, Shore ND. Enzalutamide and Quality of Life in Biochemically Recurrent Prostate Cancer. NEJM Evid. 2023 Dec;2(12):EVIDoa2300251. doi: 10.1056/EVIDoa2300251. Epub 2023 Oct 22. PMID 38320501
- [Derived] Freedland SJ, de Almeida Luz M, De Giorgi U, Gleave M, Gotto GT, Pieczonka CM, Haas GP, Kim CS, Ramirez-Backhaus M, Rannikko A, Tarazi J, Sridharan S, Sugg J, Tang Y, Tutrone RF Jr, Venugopal B, Villers A, Woo HH, Zohren F, Shore ND; EMBARK Study. Improved Outcomes with Enzalutamide in Biochemically Recurrent Prostate Cancer. N Engl J Med. 2023 Oct 19;389(16):1453-1465. doi: 10.1056/NEJMoa2303974. PMID 37851874
- [Derived] LBA02-09 EMBARK: A Phase 3 Randomized Study of Enzalutamide or Placebo Plus Leuprolide Acetate and Enzalutamide Monotherapy in High-risk Biochemically Recurrent Prostate Cancer. J Urol. 2023 Jul;210(1):224-226. doi: 10.1097/JU.0000000000003518. Epub 2023 May 2. PMID 37119051
- [Derived] Freedland SJ, De Giorgi U, Gleave M, Rosbrook B, Shen Q, Sugg J, Haas GP, Shore ND. A phase 3 randomised study of enzalutamide plus leuprolide and enzalutamide monotherapy in high-risk non-metastatic hormone-sensitive prostate cancer with rising PSA after local therapy: EMBARK study design. BMJ Open. 2021 Aug 12;11(8):e046588. doi: 10.1136/bmjopen-2020-046588. PMID 34385241

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1068 participants were enrolled and randomized to the 3 treatment groups. There were 2 participants in the enzalutamide plus leuprolide group, 4 participants in the placebo plus leuprolide group, and 1 participant in the enzalutamide monotherapy group who did not receive any study intervention.
Groups:
- Enzalutamide + Leuprolide: Participants were randomized to receive enzalutamide capsules 160 milligrams (mg)/day, plus leuprolide 22.5 mg intramuscular or subcutaneous injection once every 12 weeks from Day 1. Study treatment continued uninterrupted in the absence of disease progression until the central laboratory prostate-specific antigen (PSA) evaluation at Week 36. At week 37 study treatment was suspended for participants whose PSA values were undetectable at Week 36 and was reinitiated if subsequent PSA values increased to the threshold specified for reinitiation of study treatment. Participants with detectable PSA values at Week 36 continued treatment without suspension until permanent treatment discontinuation criteria were met.
- Placebo + Leuprolide: Participants were randomized to receive placebo capsules once daily, plus leuprolide 22.5 mg intramuscular or subcutaneous injection once every 12 weeks from Day 1. Study treatment continued uninterrupted in the absence of disease progression until the central laboratory PSA evaluation at Week 36. At week 37 study treatment was suspended for participants whose PSA values were undetectable at Week 36 and was reinitiated if subsequent PSA values increased to the threshold specified for reinitiation of study treatment. Participants with detectable PSA values at Week 36 continued treatment without suspension until permanent treatment discontinuation criteria were met.
- Enzalutamide Monotherapy: Participants were randomized to receive enzalutamide capsules 160 mg/day from Day 1. Study treatment continued uninterrupted in the absence of disease progression until the central laboratory PSA evaluation at Week 36. At week 37 study treatment was suspended for participants whose PSA values were undetectable at Week 36 and was reinitiated if subsequent PSA values increased to the threshold specified for reinitiation of study treatment. Participants with detectable PSA values at Week 36 continued treatment without suspension until permanent treatment discontinuation criteria were met.
Period: Study Treatment Phase
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Started | 355 | 358 | 355
Received Treatment | 353 | 354 | 354
Completed | 0 | 0 | 0
Not Completed | 355 | 358 | 355
Not completed — Centrally confirmed radiographic progression | 26 | 66 | 37
Not completed — PSA progression notification from sponsor | 2 | 20 | 5
Not completed — Adverse Event | 73 | 36 | 63
Not completed — Development of castration resistance | 0 | 2 | 0
Not completed — Withdrawal by Subject | 26 | 32 | 25
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — PI decision/disease progression by local conventional scan/PSA, and other miscellaneous reasons | 17 | 41 | 26
Not completed — Other | 0 | 1 | 0
Not completed — Ongoing; still in treatment phase as of primary completion date (PCD) cutoff date 31 Jan 2023 | 207 | 153 | 197
Not completed — Participants did not receive treatment. | 2 | 4 | 1
Period: Long-Term Follow-Up Phase
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Started | 148 | 205 | 158
Completed | 0 | 0 | 0
Not Completed | 148 | 205 | 158
Not completed — Ongoing; participants still in long-time follow-up phase as of the PCD cutoff date (31 January 2023) | 67 | 104 | 62
Not completed — PI decision, site closure and other miscellaneous reasons | 5 | 8 | 12
Not completed — Withdrawal by Subject | 40 | 36 | 38
Not completed — Lost to Follow-up | 3 | 3 | 4
Not completed — Death | 33 | 54 | 42

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy | Total
Number analyzed (Participants) | 353 | 354 | 354 | 1061
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (6.49) | 69.1 (7.33) | 69.1 (7.66) | 69.1 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 353 | 354 | 354 | 1061
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 0 | 5
  Asian | 26 | 26 | 26 | 78
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 16 | 16 | 15 | 47
  White | 291 | 298 | 294 | 883
  More than one race | 2 | 3 | 4 | 9
  Unknown or Not Reported | 13 | 10 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Metastasis-free Survival (MFS) Compared Between Enzalutamide Plus Leuprolide and Placebo Plus Leuprolide
Description: MFS was defined as the duration of time in months between randomization and the earliest objective evidence of radiographic progression by central imaging or death without radiographic progression, whichever occurred first. Radiographic progression for soft tissue disease was defined by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1). Radiographic progression for bone disease was defined as the appearance of 1 or more metastatic lesions on bone scan (a bone scan assesses 5 regions of the skeleton, including skull, thorax, spine, pelvis, and extremities). Confirmation with a second imaging modality (plain film, computed tomography [CT], or magnetic resonance imaging [MRI]) was to be required when bone lesions were found in a single region on the bone scan. Appearance of metastatic lesions in 2 or more of the 5 regions on a bone scan was not to require confirmation with a second imaging modality.
Time Frame: From randomization until radiographic progression or death without radiographic progression, whichever occurred first (up to Month 98 when at least 197 MFS events occurred among the 3 treatment groups)
Population: The intent-to-treat (ITT) population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide
Number analyzed (Participants) | 355 | 358
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [85.1 to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — Two-sided P-value was based on a stratified log-rank test by screening PSA, PSA doubling time, and prior hormonal therapy. Hazard ratio was based on a Cox regression model stratified by factors defined above and was relative to placebo + leuprolide with < 1 favoring enzalutamide + leuprolide; p < 0.0001, Log Rank — Statistical significance can be declared if p-value <0.05; Hazard Ratio (HR) = 0.424, 95% CI 2-sided [0.296 to 0.607]

2. Secondary Outcome: Metastasis-free Survival (MFS) Compared Between Enzalutamide Monotherapy and Placebo Plus Leuprolide
Description: MFS was defined as the duration of time in months between randomization and the earliest objective evidence of radiographic progression by central imaging or death without radiographic progression, whichever occurred first. Radiographic progression for soft tissue disease was defined by RECIST 1.1. Radiographic progression for bone disease was defined as the appearance of 1 or more metastatic lesions on bone scan (a bone scan assesses 5 regions of the skeleton, including skull, thorax, spine, pelvis, and extremities). Confirmation with a second imaging modality (plain film, CT, or MRI) was to be required when bone lesions were found in a single region on the bone scan. Appearance of metastatic lesions in 2 or more of the 5 regions on a bone scan was not to require confirmation with a second imaging modality.
Time Frame: as for outcome 1
Population: The ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Monotherapy | Placebo + Leuprolide
Number analyzed (Participants) | 355 | 358
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [85.1 to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide Monotherapy vs Placebo + Leuprolide; Test type: Other — Two-sided P-value was based on a stratified log-rank test by screening PSA, PSA doubling time, and prior hormonal therapy. Hazard ratio was based on a Cox regression model stratified by factors defined above and was relative to placebo + leuprolide with < 1 favoring enzalutamide monotherapy; p = 0.0049, Log Rank — Statistical significance can be declared if p-value <0.03; Hazard Ratio (HR) = 0.631, 95% CI 2-sided [0.456 to 0.871]

3. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as the time in months from randomization to the date of the first PSA value demonstrating progression, while participants were on study treatment, which was subsequently confirmed at least 3 weeks later. PSA progression date was defined as the date that a ≥25% increase and an absolute increase of ≥2 micrograms per liter (μg/L) (2 nanograms per milliliter [ng/mL]) above the nadir (or baseline for participants with no PSA decline by Week 25) that was confirmed by a second consecutive value at least 3 weeks later. For participants who had suspended treatment at Week 37 and later reinitiated treatment, baseline was reset as the last PSA assessment prior to or on the date of reinitiation of treatment.
Time Frame: From randomization until first PSA progression (up to Month 98)
Population: The ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — Statistical significance can be declared if p-value <0.02; Hazard Ratio (HR) = 0.068, 95% CI 2-sided [0.033 to 0.141]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Log Rank — Statistical significance can be declared if p-value <0.03; Hazard Ratio (HR) = 0.331, 95% CI 2-sided [0.226 to 0.486]

4. Secondary Outcome: Time to First Use of New Antineoplastic Therapy
Description: Time to first use of new antineoplastic therapy was defined as the time in months from randomization to first use of new antineoplastic therapy for prostate cancer.
Time Frame: From randomization until first use of new antineoplastic therapy (up to Month 98)
Population: The ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | 76.2 [71.3 to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank — Statistical significance can be declared if p-value <0.02; Hazard Ratio (HR) = 0.358, 95% CI 2-sided [0.263 to 0.488]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Log Rank — Statistical significance can be declared if p-value <0.03; Hazard Ratio (HR) = 0.540, 95% CI 2-sided [0.411 to 0.709]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time in months between randomization and death due to any cause.
Time Frame: From randomization until death due to any cause (up to Month 98 when at least 197 MFS events occurred among the 3 treatment groups)
Reporting Status: Not Posted, anticipated posting 2027-09

6. Secondary Outcome: Time to Distant Metastasis
Description: The time to distant metastasis was defined as the time in months from randomization to the earliest objective evidence of distant soft tissue metastases or metastatic bone disease by blinded independent central review (BICR).
Time Frame: From randomization until the earliest objective evidence of distant soft tissue metastases or metastatic bone disease (up to Month 98)
Population: The ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [85.1 to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.443, 95% CI 2-sided [0.284 to 0.690]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0171, Log Rank; Hazard Ratio (HR) = 0.614, 95% CI 2-sided [0.409 to 0.920]

7. Secondary Outcome: Percentage of Participants With Undetectable Prostate-specific Antigen (PSA) at 36 Weeks on Study Drug
Description: Undetectable PSA at 36 weeks was serum PSA levels <0.2 ng/mL at Week 36. Percentage of participants with undetectable PSA at 36 weeks on study drug was calculated as the number of participants with undetectable PSA at Week 36 divided by the number of participants with PSA values at Week 36, and multiplied by 100.
Time Frame: At Week 36
Population: All participants in the ITT population (randomly assigned to study treatment) who had PSA values at Week 36.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 331 | 336 | 337
Percentage of participants | 97.3 [94.9 to 98.7] | 71.4 [66.3 to 76.2] | 90.2 [86.5 to 93.2]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on a Cochran-Mantel-Haenszel test stratified by screening PSA, PSA doubling time, and prior hormonal therapy; difference of percentage of participants = 25.9, 95% CI 2-sided [20.7 to 31.0]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; difference of percentage of participants = 18.8, 95% CI 2-sided [13.0 to 24.6]

8. Secondary Outcome: Percentage of Participants Who Remained Treatment-free 2 Years After Suspension of Study Treatment at Week 37 Due to Undetectable Prostate-specific Antigen (PSA)
Description: Undetectable PSA at 36 weeks was serum PSA levels <0.2 ng/mL at Week 36. At Week 37, study treatment was suspended for participants whose PSA values were undetectable (<0.2 ng/mL) at Week 36 as determined by the central laboratory. Study treatment may have been suspended only once (at Week 37) due to undetectable PSA and was reinitiated if subsequent central laboratory PSA values increased to ≥2.0 ng/mL for participants with prior prostatectomy or ≥5.0 ng/mL for participants without prostatectomy. Percentage of participants who remained treatment-free 2 years after suspension of study treatment at Week 37 was calculated as the number of participants who remained treatment-free 2 years after suspension of study treatment at Week 37 divided by the number of participants with treatment suspension and multiplied by 100.
Time Frame: From randomization until 2 years after Week 37 (up to Month 34)
Population: All participants in the ITT population (randomly assigned to study treatment) who had treatment suspension.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 321 | 240 | 304
Percentage of participants | 34.6 [29.4 to 40.1] | 27.1 [21.6 to 33.2] | 14.1 [10.4 to 18.6]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other; p = 0.0439, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; difference of percentage of participants = 7.5, 95% CI 2-sided [-0.2 to 15.2]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other; p = 0.0004, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; difference of percentage of participants = -12.9, 95% CI 2-sided [-19.8 to -6.1]

9. Secondary Outcome: Percentage of Participants With Undetectable Prostate-specific Antigen (PSA) 2 Years After Suspension of Treatment at Week 37 Due to Undetectable PSA
Description: Undetectable PSA at 36 weeks was serum PSA levels <0.2 ng/mL at Week 36. At Week 37, study treatment was suspended for participants whose PSA values were undetectable (<0.2 ng/mL) at Week 36 as determined by the central laboratory. Study treatment may have been suspended only once (at Week 37) due to undetectable PSA and was reinitiated if subsequent central laboratory PSA values increased to ≥2.0 ng/mL for participants with prior prostatectomy or ≥5.0 ng/mL for participants without prostatectomy. Percentage of participants with undetectable PSA 2 years after suspension of treatment at Week 37 due to undetectable PSA was calculated as the number of participants with undetectable PSA 2 years after suspension of treatment at Week 37 due to undetectable PSA divided by the number of participants with treatment suspension and multiplied by 100.
Time Frame: From randomization until 2 years after Week 37 (up to Month 34)
Population: All participants in the ITT population (randomly assigned to study treatment) who had treatment suspension.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 321 | 240 | 304
Percentage of participants | 16.8 [12.9 to 21.4] | 9.6 [6.2 to 14.0] | 4.6 [2.5 to 7.6]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other; p = 0.0089, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; difference of percentage of participants = 7.2, 95% CI 2-sided [1.7 to 12.8]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other; p = 0.0326, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; difference of percentage of participants = -5.0, 95% CI 2-sided [-9.4 to -0.6]

10. Secondary Outcome: Time to Resumption of Any Hormonal Therapy Following Suspension at Week 37 Due to Undetectable Prostate-specific Antigen (PSA)
Description: Undetectable PSA at 36 weeks was serum PSA levels <0.2 ng/mL at Week 36. At Week 37, study treatment was suspended for participants whose PSA values were undetectable (<0.2 ng/mL) at Week 36 as determined by the central laboratory. Study treatment may have been suspended only once (at Week 37) due to undetectable PSA and was reinitiated if subsequent central laboratory PSA values increased to ≥2.0 ng/mL for participants with prior prostatectomy or ≥5.0 ng/mL for participants without prostatectomy. The time to resumption of any hormonal therapy following suspension at Week 37 due to undetectable PSA was defined as the time in months between the date of treatment suspension at Week 37 due to undetectable PSA and the date that hormonal therapy was restarted.
Time Frame: From treatment suspension at Week 37 until resumption of any hormonal therapy (up to Month 98)
Population: All participants in the ITT population (randomly assigned to study treatment) who had treatment suspension.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 321 | 240 | 304
Months | 19.6 [17.2 to 22.3] | 16.8 [14.3 to 17.1] | 10.5 [8.9 to 11.5]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.577 to 0.834]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 1.655, 95% CI 2-sided [1.381 to 1.984]

11. Secondary Outcome: Time to Castration Resistance
Description: Time to castration resistance applied only to participants receiving leuprolide treatment and was defined as the time in months from randomization to the first occurrence of radiographic disease progression by BICR, PSA progression or symptomatic skeletal event (SSE) whichever occurred first with castrate levels of testosterone (<50 ng/dL).
Time Frame: From randomization to the first occurrence of radiographic disease progression, PSA progression or SSE, whichever occurred first with castrate levels of testosterone (up to Month 98)
Population: The ITT population was used for analysis, and it included all participants randomly assigned to receive leuprolide treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide
Number analyzed (Participants) | 355 | 358
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.090, 95% CI 2-sided [0.051 to 0.157]

12. Secondary Outcome: Time to Symptomatic Progression
Description: Time to symptomatic progression was defined as the time in months from randomization to development of a skeletal-related event, worsening of disease-related symptoms requiring initiation of a new antineoplastic therapy, or development of adverse events (AEs) and clinically significant signs and/or symptoms due to loco-regional tumor progression requiring opiate use, surgical intervention or radiation therapy, whichever occurred first.
Time Frame: From randomization until the first development of events defined as symptomatic progression (up to Month 98)
Population: ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | 63.8 [56.4 to 74.9] | NA [83.6 to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.546, 95% CI 2-sided [0.427 to 0.699]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.619, 95% CI 2-sided [0.488 to 0.785]

13. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: Time to first symptomatic skeletal event was defined as the time in months from randomization to use of radiation therapy (external beam radiation therapy or radionuclides) or surgery to bone for prostate cancer, findings of clinically apparent pathologic bone fracture or of spinal cord compression, or new use of opiate and/or systemic antineoplastic therapy due to bone pain collected in the SSE case report form (CRF), whichever occurred first.
Time Frame: From randomization until the first development of events defined as SSE (up to Month 98)
Population: ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events. | NA [NA to NA] — NA indicates not estimable due to small number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.261, 95% CI 2-sided [0.125 to 0.548]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0057, Log Rank; Hazard Ratio (HR) = 0.423, 95% CI 2-sided [0.226 to 0.794]

14. Secondary Outcome: Time From Randomization to Onset of Clinically Relevant Pain Progression, Defined as a 2-point or Greater Increase From Baseline in the Brief Pain Inventory-Short Form (BPI-SF) Question 3 Score
Description: Time to clinically relevant pain progression was defined as the time from randomization to onset of pain progression, where clinically relevant pain progression was defined as a 2-point or greater increase from baseline in the BPI-SF question 3 score. BPI-SF is a self-administered questionnaire containing 9 main questions related to pain and analgesic medication use, where question 3 (paraphrased) is "On a scale of 0 [no pain] to 10 [pain as bad as you can imagine], please rate your pain at its worst in the last 24 hours" with higher score indicating worse pain.
Time Frame: From randomization until a 2-point or greater increase from baseline in the BPI-SF question 3 score (up to Month 98)
Population: ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | 13.9 [11.9 to 19.4] | 19.4 [13.8 to 24.9] | 16.6 [12.3 to 19.4]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.4321, Log Rank; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.894 to 1.301]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.3702, Log Rank; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.904 to 1.314]

15. Secondary Outcome: Time From Randomization to First Assessment With at Least a 10-point Decline (Deterioration) From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Total Score
Description: Time to first deterioration of the FACT-P total score was defined as the time from randomization to first assessment with at least a 10-point decrease from baseline in the FACT-P total score. FACT-P total score is based on subscale scores of physical, social/family, emotional, and functional well-being, as well as 12 site-specific items to assess prostate-related symptoms, ranging 0-156, with higher score representing better quality of life.
Time Frame: From randomization to first assessment with at least a 10-point decrease from baseline in the FACT-P total score (up to Month 98)
Population: ITT population was used for analysis, and it included all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
Number analyzed (Participants) | 355 | 358 | 355
Months | 8.3 [5.7 to 11.1] | 11.1 [8.3 to 14.0] | 8.4 [5.8 to 13.0]
Statistical Analysis 1: Comparison: Enzalutamide + Leuprolide vs Placebo + Leuprolide; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1567, Log Rank; Hazard Ratio (HR) = 1.138, 95% CI 2-sided [0.954 to 1.357]
Statistical Analysis 2: Comparison: Placebo + Leuprolide vs Enzalutamide Monotherapy; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0855, Log Rank; Hazard Ratio (HR) = 1.168, 95% CI 2-sided [0.981 to 1.391]

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (All-causality) During On-treatment Period, Modified Treatment Period, and Treatment Reinitiation Period - at PCD Cut-off Date of 31 January 2023
Description: An AE was any untoward medical occurrence (eg, sign, symptom, illness, disease or injury) in a participant administered study drug or other protocol-imposed intervention, regardless of attribution. TEAEs were those events with onset dates occurring during the on-treatment period for the first time. On-treatment period was the time from the date of first dose of study treatment through a minimum of 30 days after last dose of study treatment, or the start day of new antineoplastic drug therapy minus 1 day. Modified TEAEs (mTEAEs) were AEs that occurred during the modified treatment period (events occurring or worsening during the treatment suspension period after 30 days of last dose prior to treatment suspension were excluded). Reinitiated TEAEs (rTEAEs) were AEs that occurred with a start date during the dosing period after suspension and reinitiation of study treatment as defined by the reinitiation treatment period.
Time Frame: From first dose of study drug to the last dose + 30 days, or the day before initiation of a new antineoplastic treatment (up to Month 98)
Reporting Status: Not Posted, anticipated posting 2027-09

17. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment-emergent Adverse Events (TEAEs) (All-causality) - at PCD Cut-off Date of 31 January 2023
Description: An AE was any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a participant administered study drug or other protocol-imposed intervention, regardless of attribution. TEAEs were those events with onset dates occurring during the on-treatment period for the first time. On-treatment period was defined as the time from the date of first dose of study treatment through a minimum of 30 days after last dose of study treatment, or the start day of new antineoplastic drug therapy minus 1 day. The severity of all TEAEs was evaluated by the investigator based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (potentially life-threatening) and grade 5 (death related to AE).
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

18. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (Treatment-related) During On-treatment Period, Modified Treatment Period, and Treatment Reinitiation Period - at PCD Cut-off Date of 31 January 2023
Description: An AE was any untoward medical occurrence (eg, sign, symptom, illness, disease or injury) in a participant administered study drug or other protocol-imposed intervention, regardless of attribution. TEAEs were those with onset dates occurring during the on-treatment period for the first time. On-treatment period was the time from date of first dose of study treatment through at least 30 days after last dose of study treatment or start day of new antineoplastic drug therapy minus 1 day. Treatment-related TEAEs were TEAEs attributed to study drug (enzalutamide, placebo or leuprolide). mTEAEs were AEs that occurred during the modified treatment period (events occurring or worsening during the treatment suspension period after 30 days of last dose prior to treatment suspension were excluded). rTEAEs were AEs that occurred with a start date during the dosing period after suspension and reinitiation of study treatment (reinitiation treatment period).
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

19. Secondary Outcome: Number of Participants With SAEs (All-causality) During On-treatment Period, Modified Treatment Period and Treatment Reinitiation Period and SAEs (Treatment-related) During On-treatment period-at PCD Cut-off 31 Jan 2023
Description: An AE was any untoward medical occurrence in a participant administered study drug/other protocol-imposed intervention regardless of attribution. SAEs were AEs resulting in any of the following outcomes/deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent/significant disability/incapacity; congenital anomaly. On-treatment period was time from first dose date of study treatment through ≥30 days after last dose of study treatment or start day of new antineoplastic drug therapy -1 day. mSAEs were SAEs occurring during modified treatment period (events occurring/worsening during treatment suspension period after 30 days of last dose prior to treatment suspension were excluded). rSAEs were SAEs occurring with a start date during the dosing period after suspension and reinitiation of study treatment. Treatment-related SAEs were attributed to any study drug.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Enzalutamide or Placebo Discontinuation - at PCD Cut-off Date of 31 January 2023
Description: An AE was any untoward medical occurrence (eg, sign, symptom, illness, disease or injury) in a participant administered study drug or other protocol-imposed intervention, regardless of attribution. TEAEs were those events with onset dates occurring during the on-treatment period for the first time. On-treatment period was the time from the date of first dose of study treatment through a minimum of 30 days after last dose of study treatment, or the start day of new antineoplastic drug therapy minus 1 day.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

21. Secondary Outcome: Number of Participants With Shifts From Grade ≤2 at Baseline to Grade 3 or Grade 4 Post-baseline in Hematology Laboratory Test Values - at PCD Cut-off Date of 31 January 2023
Description: Participants who experienced hematology laboratory test abnormalities were summarized according to worst toxicity grade observed for each hematology laboratory test. Hematology laboratory abnormalities were graded according to CTCAE version 4.03 (Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death). This outcome measure calculated the number of participants with hematology laboratory abnormalities that were shifted from ≤Grade 2 at baseline to Grade 3 and Grade 4 post-baseline for the following parameters: hemoglobin, leukocytes, lymphocytes, neutrophils, platelets.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

22. Secondary Outcome: Number of Participants With Shifts From Grade ≤2 at Baseline to Grade 3 or Grade 4 Post-baseline in Chemistry Laboratory Test Values - at PCD Cut-off Date of 31 January 2023
Description: Participants who experienced chemistry laboratory test abnormalities were summarized according to worst toxicity grade observed for each chemistry laboratory test. Chemistry laboratory abnormalities were graded according to CTCAE version 4.03 (Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death). This outcome measure calculated the number of participants with chemistry laboratory abnormalities that were shifted from ≤Grade 2 at baseline to Grade 3 and Grade 4 post-baseline for the following parameters: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, calcium, creatine kinase, glucose, magnesium, phosphate, potassium, sodium.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

23. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs - at PCD Cut-off Date of 31 January 2023
Description: Participants with potentially clinically significant abnormalities in vital signs were summarized for the following parameters: systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR). Potentially clinically significant abnormalities were defined as (1) SBP (mmHg): >180 and increase from baseline >40; <90 and decrease from baseline >30; final visit or 2 consecutive visits change from baseline (CFB) ≥10, ≥15, ≥20; final visit or most extreme result ≥140, ≥180, ≥140 and ≥20 CFB, ≥180 and ≥20 CFB; (2) DBP (mmHg): >105 and increase from baseline >30; <50 and decrease from baseline >20; final visit or 2 consecutive visits CFB ≥5, ≥10, ≥15; final visit or most extreme result ≥90, ≥105, ≥90 and ≥15 CFB, ≥105 and ≥15 CFB; (3) HR (bpm): >120 and increase from baseline >30; <50 and decrease from baseline >20.
Time Frame: as for outcome 16
Reporting Status: Not Posted, anticipated posting 2027-09

ADVERSE EVENTS:
Time Frame: The treatment-emergent safety reporting period was from the first dose of study treatment on Day 1 through a minimum of 30 days after the last dose of study treatment, or the start day of new antineoplastic drug therapy minus 1 day (up to 98 months). For all-cause mortality, deaths as of the PCD data cutoff include deaths occuring during and after the treatment-emergent safety reporting period.
Description: For all-cause mortality, ITT population was used for analysis, which included all participants randomly assigned to treatment. For serious adverse events and other adverse events, safety population was used for analysis, which included all randomized participants who received at least 1 dose of any study treatment.
Arm/Group | Enzalutamide + Leuprolide | Placebo + Leuprolide | Enzalutamide Monotherapy
All-Cause Mortality (participants affected / at risk) | 33/355 | 55/358 | 42/355
Serious Adverse Events (participants affected / at risk) | 123/353 | 112/354 | 131/354
Other Adverse Events (participants affected / at risk) | 339/353 | 341/354 | 345/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide + Leuprolide (N=353) | Placebo + Leuprolide (N=354) | Enzalutamide Monotherapy (N=354)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic embolism (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 4 | 3
Angina pectoris (Cardiac disorders) | 3 | 0 | 4
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 2 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1 | 8
Coronary artery occlusion (Cardiac disorders) | 2 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 3
Dressler's syndrome (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 2 | 5
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Alcohol interaction (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 2 | 0
Condition aggravated (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 3
Disease progression (General disorders) | 2 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1
Mesenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 4
Volvulus of small bowel (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0
Ocular surface stem cell transplant rejection (Immune system disorders) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Brucellosis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 4 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 1
Focal peritonitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1
Large intestine infection (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 2
Penile infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 8 | 4 | 5
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Pyelitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 4 | 4 | 6
Skin infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 5
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 2 | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 1 | 0
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Biopsy lymph gland normal (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood osmolarity decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 3 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-secretory adenoma of pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 3 | 3 | 2
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 3 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Post stroke epilepsy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 3 | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 9 | 4 | 2
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 2 | 2
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 1
Device loosening (Product Issues) | 1 | 0 | 0
Device material issue (Product Issues) | 0 | 1 | 1
Device occlusion (Product Issues) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 2
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 4
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 2
Bladder stenosis (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 8 | 4 | 8
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 3
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 3 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 5
Urinary retention (Renal and urinary disorders) | 1 | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Immobile (Social circumstances) | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Dry gangrene (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide + Leuprolide (N=353) | Placebo + Leuprolide (N=354) | Enzalutamide Monotherapy (N=354)
Anaemia (Blood and lymphatic system disorders) | 24 | 11 | 17
Cataract (Eye disorders) | 17 | 20 | 22
Asthenia (General disorders) | 39 | 21 | 39
Fatigue (General disorders) | 151 | 116 | 165
Oedema peripheral (General disorders) | 27 | 36 | 31
Constipation (Gastrointestinal disorders) | 46 | 31 | 33
Diarrhoea (Gastrointestinal disorders) | 49 | 30 | 46
Dyspepsia (Gastrointestinal disorders) | 7 | 9 | 20
Nausea (Gastrointestinal disorders) | 42 | 29 | 53
Bronchitis (Infections and infestations) | 19 | 12 | 10
COVID-19 (Infections and infestations) | 25 | 34 | 42
Nasopharyngitis (Infections and infestations) | 25 | 22 | 31
Upper respiratory tract infection (Infections and infestations) | 21 | 25 | 22
Urinary tract infection (Infections and infestations) | 26 | 25 | 33
Fall (Injury, poisoning and procedural complications) | 72 | 50 | 52
Overdose (Injury, poisoning and procedural complications) | 10 | 12 | 18
Rib fracture (Injury, poisoning and procedural complications) | 29 | 23 | 18
Weight decreased (Investigations) | 24 | 12 | 39
Weight increased (Investigations) | 27 | 30 | 17
Decreased appetite (Metabolism and nutrition disorders) | 27 | 15 | 32
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 17 | 18 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 97 | 74 | 80
Arthritis (Musculoskeletal and connective tissue disorders) | 14 | 13 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 54 | 61
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 19 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 16 | 18 | 14
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 13 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 39 | 36 | 40
Dizziness (Nervous system disorders) | 39 | 37 | 41
Headache (Nervous system disorders) | 39 | 32 | 41
Memory impairment (Nervous system disorders) | 26 | 12 | 21
Anxiety (Psychiatric disorders) | 18 | 11 | 18
Depression (Psychiatric disorders) | 21 | 20 | 21
Insomnia (Psychiatric disorders) | 42 | 37 | 25
Dysuria (Renal and urinary disorders) | 12 | 18 | 10
Haematuria (Renal and urinary disorders) | 38 | 41 | 43
Nocturia (Renal and urinary disorders) | 26 | 16 | 9
Pollakiuria (Renal and urinary disorders) | 30 | 30 | 27
Urinary incontinence (Renal and urinary disorders) | 34 | 28 | 32
Breast pain (Reproductive system and breast disorders) | 4 | 3 | 25
Breast tenderness (Reproductive system and breast disorders) | 5 | 4 | 51
Gynaecomastia (Reproductive system and breast disorders) | 29 | 32 | 159
Nipple pain (Reproductive system and breast disorders) | 11 | 4 | 54
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 24 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 23 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 2 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 4 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 10 | 17
Rash (Skin and subcutaneous tissue disorders) | 22 | 23 | 22
Hot flush (Vascular disorders) | 243 | 203 | 77
Hypertension (Vascular disorders) | 82 | 69 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02319837/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02319837/SAP_001.pdf